CLINICAL TRIAL: NCT06088108
Title: Age and Sex Differences in the Metabolic Response to Exercise
Brief Title: Metabolic Responses to Exercise and Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University of East London (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Metabex
Record Dates: First submitted 2023-10-04; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Exercise; Metabolism
Keywords: Exercise; Metabolism; Recovery; Metabolomics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Study participants are asked to undertake the Cornell treadmill exercise protocol which they complete to voluntary exhaustion.
  Interventions: Device: Cornell treadmill exercise protocol

INTERVENTIONS:
Device: Cornell treadmill exercise protocol — Study participants are asked to undertake the Cornell treadmill exercise protocol which they complete to voluntary exhaustion.

SUMMARY:
Exercise benefits health through diverse metabolic processes and is central to healthy ageing. However, intense exercise also challenges the body, causing cellular damage that must be repaired. This means that we need to identify the level of exercise that can optimise health, and this level might potentially differ by age and sex. Our research aims to tackle this question, by studying the metabolic responses of the body both to exercise and during the subsequent recovery in 48 healthy and active participants between the ages of 8-10, 23-27 and 53-57.

Participants will complete an inclusion questionnaire and, if eligible, be invited to visit the exercise laboratory 4-5-hours. We will collect questionnaire data and body measurements before participants undertake exercise on a treadmill. Biological samples (blood from adults only and saliva from everyone) will be collected at three time points (before, right after and one hour after exercise).

DETAILED DESCRIPTION:
Before taking part, participants will be asked to complete an online inclusion questionnaire where the investigators will ask some questions about their health status, weight status, lifestyle, and medications to confirm that the participants are eligible and that it is safe for the participants to participate in the study. The investigators will record their consent electronically at this stage. If the participants are eligible and decide to take part in the study, the investigators will ask the participants to record their consent in writing before proceeding further.

The in-person part of the study will take place at the University Of East London SportsDock (4-6 University Way, London E16 2RD) and last 4-5 hours. No breakfast or coffee/tea should be consumed on the day of the visit, but the investigators will offer the participants breakfast. The participants will also need to not have had any alcohol, recreational drugs, or exercise for 24 hours.

On the day, the investigators will first measure their resting heart rate and blood pressure, collect body measurements (weight, height, waist circumference, hip circumference), and measure their body composition. The last thing the investigators will do before breakfast is to collect some samples. The investigators will collect two separate saliva samples using synthetic cotton swabs. After this, the investigators will collect a blood sample by venepuncture ("needle prick") from the adults only. This first part of the study will take 45-60 minutes.

Along with breakfast, the investigators will ask the participants to consume a dose of deuterium-labelled water: an odourless, tasteless, and safe water that will allow us to measure their total body water content. The investigators will also ask the participants to complete two short questionnaires assessing their mood, appetite, feeling of tiredness as well as verbal learning. This part will take approximately 30 minutes.

The researcher will then help the participants familiarise with the treadmill and associated equipment. The participants will wear a chest strap under their clothes and a special face mask which will be held in place by a head strap. These will measure their heart rate and everything the participants breathe in and out throughout the exercise challenge, respectively. The treadmill will start slowly to help the participants warm up and familiarise with the feeling of walking on it. After 2 minutes, the exercise challenge will begin. This will last for approximately 20 minutes, during which the treadmill will increase the speed and/or the incline every 2 minutes. It will feel like the participants are walking more briskly and more uphill, but it will not be too fast. The researcher will encourage the participants to complete the exercise challenge, as this will get the best response from their metabolism and give us the most accurate results. The participants will be able to stop the treadmill if the participants feel too exhausted to continue, feel faint or develop chest pain.

Right after the participants complete the exercise challenge, the investigators will collect a saliva sample using a synthetic cotton swab and a blood sample by venepuncture (adults only). The investigators will then ask the participants to complete the same two short questionnaires as before. This part will take approximately 30 minutes.

Finally, the researcher will allow the participants to relax and rest for about an hour. The investigators will then collect the last saliva samples using synthetic cotton swabs and blood samples by venepuncture (adults only). The participants will then complete the last iteration of the two short questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 8-10, 23-27 or 53-57
2. Considered healthy without a disease, disability or other condition that would impair participation in physical activity.
3. Considered active.
4. A body mass index within the ranges of 19 to 24.5 (adults) or the 2nd and 99th percentile (children)

Exclusion Criteria:

1. Outside required age brackets
2. Having a disease, disability or other condition that would impair participation in physical activity.
3. Having an implanted cardiac pacemaker, defibrillator, or other electronic medical devices.
4. Receiving prescription medication one or more days every week over the past 3 months (some medications are permitted).
5. Related by blood to another participant.
6. Not willing at the time of recruitment to undergo blood sampling (adults only).
7. Pregnancy/breastfeeding (adults only).
8. Being a professional athlete.
9. Not being physically active.
10. Being a shift worker (night shift work for three or more days per week on more than two occasions in the six months before the visit day; adults only).
11. Recent weight loss of more than 5% of weight in the last 6 months.
12. Having a body mass index outside the range of 19 to 24.5 (adults) or outside the 2nd and 99th percentile (children)
13. Smoking/vaping.
14. Alcohol intake above a UK National Health Service (NHS) questionnaire cut-off.
15. Regular use of recreational drugs.
16. Not having reached menopause (for women aged 53-57 only).

Ages: 8 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of molecules relating to energy metabolism using targeted liquid chromatography-mass spectrometry assays | At baseline, immediately after exercise and one hour after exercise
  Concentrations of metabolites measured in plasma and saliva at baseline, immediately after exercise and one hour after exercise using targeted liquid chromatography-mass spectrometry (LCMS) assays. These include amine, ion-pairing, lipid, fatty acid, acylcarnitine and oxylipin assays.

SECONDARY OUTCOMES:
Concentrations of hormones relating to life history functions using different assays | At baseline, immediately after exercise and one hour after exercise
  Concentrations of hormones measured in plasma or saliva at baseline, immediately after exercise and one hour after exercise using hormone assays. These hormone assays relate to the four life history functions, maintenance, defence, reproduction and growth. The following assays will be used: Bacteria killing and haemolytic complement assays in plasma to assess resistance to infection, total antioxidant capacity and malondialdehyde assays in plasma to assess oxidative stress, cortisol in saliva to assess stress response, interleukin-6 in saliva to assess inflammation, insulin growth factor and growth hormone assays in saliva to assess growth, oestradiol and testosterone in saliva to assess reproduction, as well as leptin, adiponectin and insulin in saliva to assess energy stores.
Total body water measurement | Saliva collection before and 4 hours following consumption of deuterium
  Total body water using the doubly-labelled water method which involves collection of saliva before and 4 hours after consuming a dose of deuterium
Verbal memory | Baseline, immediately after exercise and one hour after exercise
  Verbal memory assessment using the Rey Auditory Verbal Learning Test (RAVLT)
Measurement of stress, mood, appetite perception, and the desire to eat different types of food | Before breakfast, after breakfast as well as 15, 30, 45 and 60 minutes after exercise
  Assessment of stress, mood, appetite perception, and the desire to eat different types of food using a visual analogue scale published by Stubbs et al, 2000 and adapted online before breakfast, after breakfast as well as 15, 30, 45 and 60 minutes after exercise. This instrument incorporates a straight line in between two opposing statements defined as 'very little' to 'very much'. Participants are asked to mark a point in relation to their feelings at that moment.
  Stubbs, R. J., Hughes, D. A., Johnstone, A. M., Rowley, E., Reid, C., Elia, M., et al. (2000). The use of visual analogue scales to assess motivation to eat in human subjects: A review of their reliability and validity with an evaluation of new hand-held computerized systems for temporal tracking of appetite ratings. British Journal of Nutrition, 84, 405e415.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wells, Professor, Principal Investigator — University College, London
Locations (1):
- University of East London SportsDock, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers will have access to fully anonymised data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It will be available on UCL's repository from March 2025 onwards.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT06088108/ICF_000.pdf